CLINICAL TRIAL: NCT01757743
Title: Protein Distribution and Colloid Osmotic Pressure in Children With Volume and Pressure Loading Due to Congenital Heart Defects
Brief Title: Fluid Balance During Closure of Atrial Septal Defect
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Marianne Indrebo, MD Research fellow, Oslo University Hospital
Other Study IDs: 063.09
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Heart Defects,Congenital; Heart Septal Defects, Atrial
Keywords: Heart Septal Defects, Atrial; Oedema formation
MeSH Terms: conditions — Heart Defects, Congenital; Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Interstitial fluid Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Interventional closure: Interventional catheterization closure
- Open Heart Surgery: Surgery for Atrial septal defect

SUMMARY:
This project will evaluate fluid balance and oedema formation in children with the same congenital heart disease (Atrial Septal Defect) who will either go through heart surgery with the use of Cardio Pulmonary Bypass and hypothermia or through interventional catheterization. The investigators will measure interstitial colloid osmotic pressure, distribution of proteins and cytokines. The study hypothesis is that "Oedema developed during heart surgery is caused by reduced colloid osmotic pressure gradient through the capillary membrane".

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of Atrial Septal Defect scheduled for closure
* Informed consent

Exclusion Criteria:

* Renal failure,
* liver failure,
* coexisting cardiac malformations

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Atrial Septal Defect scheduled for interventional closure with device or surgical repair
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Interstitial colloid osmotic pressure | During surgery or interventional closure

CONTACTS AND LOCATIONS:
Overall Officials: Marianne M Indrebo, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided